CLINICAL TRIAL: NCT03121859
Title: Does The Use Of Analgesic Current Therapies Increase The Effectiveness Of Neck Stabilization Exercises For Improving Pain, Disability, Mood, And Quality Of Life In Chronic Neck Pain? A Randomized, Controlled, Single-Blind Study
Brief Title: Analgesic Current Therapies for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Yeşil (Other)
Responsible Party: Sponsor-Investigator, Hilal Yeşil, Assist Prof, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-SHHY
Record Dates: First submitted 2017-04-10; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Chronic Neck Pain
Keywords: TENS; interferential current therapy; Chronic neck pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neck stabilization exercise (Active Comparator): The patients who had only neck stabilization exercise
  Interventions: Other: Neck stabilization exercise
- TENS+ neck stabilization exercise (Active Comparator): The patients who had both TENS and neck stabilization exercise
  Interventions: Other: Neck stabilization exercise; Other: TENS
- IFC+ neck stabilization exercise (Active Comparator): The patients who had both interferential current therapy and neck stabilization exercise
  Interventions: Other: Neck stabilization exercise; Other: IFC

INTERVENTIONS:
Other: Neck stabilization exercise — Exercise
Other: TENS — Transcutaneous electrical nerve stimulation (TENS)
  Arms: TENS+ neck stabilization exercise
Other: IFC — Interferential current therapy(IFC)
  Arms: IFC+ neck stabilization exercise

SUMMARY:
Does the use of analgesic current therapies increase the effectiveness of neck stabilization exercises for improving pain, disability, mood, and quality of life in chronic neck pain? a randomized, controlled, single-blind study

DETAILED DESCRIPTION:
Analgesic therapies; such as interferential current (IFC) and transcutaneous electrical nerve stimulation (TENS) have been applied solo or combined with exercise for management of neck pain (NP), however, the efficacy of these combinations are unclear. In this study, our objective were to determine if TENS or IFC increase the effectiveness of neck stabilization exercises on pain, disability, mood, and quality of life for chronic NP. 81 patients with chronic NP were included in the study. Patients were randomly assigned into 3 groups; Group I: neck stabilization exercise, Group II: TENS+ neck stabilization exercise and Group III: IFC+ neck stabilization exercise. Patients' pain levels (visual analogue scale (VAS)), quality of life (short form- 36), mood (Beck depression inventory (BDI)), levels of disability (Neck Pain and Disability Index) and the need for analgesics were evaluated prior to treatment, at 6th and 12th week follow-up. All participants had group exercise accompanied by a physiotherapist for 3 weeks and an additional 3 weeks of home exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Both genders between 20-50 years, had chronic neck pain

Exclusion Criteria: Having disc hernia that causes neurological deficit

* Having malignity,
* Having neck pain secondary neurological or vascular disease.
* Pregnancy
* Having psychiatric disease
* Having arthritic disease
* Having any contraindication for electrotherapy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline VAS (Visual analog scale) at 6th and 12th weeks | Up to12 weeks
  The patients were asked to make an assessment of their pain between 0 (no pain) and 10 (severe pain).

SECONDARY OUTCOMES:
Change from baseline quality of life (short form- 36) at 6th and 12th weeks | Up to 12 weeks
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health.
Change from baseline Beck depression inventory (BDI) at 6th and 12th weeks | Up to 12 weeks
  The Beck Depression Inventory (BDI); was used to assess the depression levels of the patients. The BDI evaluates 21 symptoms of depression. These symptoms deal with emotions, behavioral changes, and somatic symptoms. Each symptom is rated on a 4-point intensity scale. Higher scores indicate more severe depression
Change from baseline Neck Pain and Disability Index at 6th and 12th weeks | Up to 12 weeks
  The questionnaire consists of 20 items and measures neck movements, pain intensity, effect of neck pain on emotion factors, and interference with daily life activities. Each section is scored on a 0-5 rating scale and total score ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal Yesil, Afyonkarahisar, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No